CLINICAL TRIAL: NCT07135232
Title: The Effects of Resistance Training and a Sarmentosin - L-theanine Supplement on Perimenopausal Symptoms and Musculoskeletal Health: A Randomised Controlled Trial
Brief Title: The Effects of Resistance Training and a Plant-Based Supplement on Perimenopausal Symptoms and Muscle Health.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Leeds Beckett University (Other)
Responsible Party: Principal Investigator, Harriet Cannell, Doctoral Researcher, Leeds Beckett University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AM004156
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Perimenopause; Menopause
Keywords: Mood; Depression; Cognition; Resistance Training; Sarmentosin - L-theanine; Bioactive supplement; perimenopause symptoms; menopause; lifestyle; muscle; health; exercise; perimenopause; symptoms; hot flashes; vasomotor; anxiety; stress
MeSH Terms: conditions — Depression; Motor Activity; Hot Flashes; Anxiety Disorders | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Masking will only be applied to supplement allocation. All parties will be aware of their exercise allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo Supplement Only (Placebo Comparator): One placebo capsule to be consumed by participants daily
  Interventions: Dietary Supplement: Placebo Supplement
- Placebo Supplement and Resistance Training (Experimental): Participants will consume one placebo supplement daily, and perform structured resistance training three times per week.
  Interventions: Other: Resistance Training; Dietary Supplement: Placebo Supplement
- Active Supplement Only (Experimental): Participants will consume one capsule of the Sarmentosin - L-theanine supplement daily.
  Interventions: Dietary Supplement: Sarmentosin - L- theanine
- Active Supplement and Resistance Training (Experimental): Participants will consume one capsule of the Sarmentosin - L-theanine supplement daily and perform structured resistance training three times per week.
  Interventions: Dietary Supplement: Sarmentosin - L- theanine; Other: Resistance Training

INTERVENTIONS:
Dietary Supplement: Sarmentosin - L- theanine — A capsule containing 20 mg of Sarmentosin and 400mg of L-theanine
  Arms: Active Supplement Only; Active Supplement and Resistance Training
Other: Resistance Training — Home-based Resistance training. Exercises will target the lower and upper body and utilise body weight, resistance bands, dumbbells and push-up handles.
  Other Names: Strength Training; Resistance Exercise; Strength Exercise
  Arms: Active Supplement and Resistance Training; Placebo Supplement and Resistance Training
Dietary Supplement: Placebo Supplement — Capsule matched for taste and appearance, without any active ingredients.
  Arms: Placebo Supplement Only; Placebo Supplement and Resistance Training

SUMMARY:
The aim of this clinical trial is to determine if resistance training and a newly developed plant-based nutritional supplement can improve the symptoms and musculoskeletal health of perimenopausal women.

The main questions it aims to evaluate are:

1. Can resistance training and the nutritional supplement - both independently and in combination - improve perimenopausal symptoms (e.g. cognition, mood, sleep) and musculoskeletal outcomes (e.g. strength, muscle mass)?
2. What are the acute effects of the nutritional supplement on cognitive function and mood in perimenopausal women, and is this response altered following long-term intake (12 weeks)?
3. What mechanisms may be contributing to the results?

Participants will be split into four groups to allow the researchers to answer the above questions. These are:

1. The nutritional supplement + resistance training
2. The nutritional supplement only
3. The placebo supplement (A look alike capsule that contains no active ingredients) and resistance training
4. The Placebo supplement only.

Participants will:

* Take their allocated supplement daily and perform home-based strength exercise 3 times per week (for exercise groups), for 12 weeks.
* Attend the laboratory at the beginning and end of the 12 weeks to assess cognitive function and mood following acute intake of the supplement.
* Attend the laboratory every 4 weeks during the 12 week period, for assessment of cognitive function, symptom severity and muscle health.
* Provide a blood sample at each visit for assessment of mechanistic pathways.

ELIGIBILITY:
Inclusion criteria

1. Perimenopausal women between 40 - 55 years
2. Not currently engaging in consistent structured resistance training (defined as >3 resistance training sessions per week for 4 consecutive weeks, in the past six months).
3. Not on any HRT or hormonal contraception for at least one year before initiation of the study.
4. Able to attend laboratory visits and commit to the intervention schedule for 6 months.
5. Willing to provide blood samples
6. Not regularly consuming any dietary supplements containing concentrated sarmentosin, L-theanine or other compounds that may interfere with the study intervention.
7. Willing to limit dietary intake of Sarmentosin (e.g. Blackcurrant) and L-theanine (e.g. green tea/ black tea).
8. Willing and able to provide written informed consent

Exclusion criteria

1. Diagnosed cardiovascular disease (CVD), uncontrolled hypertension (>160/100 mmHg), or other conditions that prevent safe exercise participation.
2. Clinically diagnosed mental health disorders (e.g., bipolar disorder, schizophrenia, severe depression requiring medication adjustment within the last 6 months).
3. Neurological conditions affecting cognitive function (e.g., Parkinson's disease, multiple sclerosis, epilepsy).
4. Endocrine disorders that could impact hormonal fluctuations or metabolism (e.g., uncontrolled diabetes, thyroid dysfunction).
5. History of major musculoskeletal injuries (e.g., fractures, joint replacement) within the past 6 months
6. Regular use of medications that could interfere with study outcomes, including antidepressants, corticosteroids, beta-blockers.
7. Obesity (BMI >30 or for South Asian Ethinicity BMI> 27.5)
8. Food allergy or intolerance to study products.
9. Use of illicit drugs.
10. Alcohol intake exceeding the government guidelines of 14 standard units per week (Equivalent of 6 standard drinks).
11. Pregnant or planning to conceive during the trial.
12. High habitual caffeine intake (>400 mg/day which is approximately 4-5 cups of coffee)

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must have been assigned female at birth.
Enrollment: 72 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Depressive Symptom Score at week 4 | Week 4
  Assessed using the depressive sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe depressive symptoms.
Depressive Symptom Score at Week 8 | Week 8
  Assessed using the depressive sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe depressive symptoms.
Depressive Symptom Score at Week 12 | Week 12
  Assessed using the depressive sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe depressive symptoms.
Change in Sustained Attention Pre- to Post-Supplement Intake at Week 1 | Pre- to 1 hour post- supplement intake at week 1 of the intervention.
  Assessed as the signal detection measure of a subject's sensitivity to the target sequence (A') during the Cambridge Neuropsychological Test Automated Battery rapid visual information processing test.
Change in Sustained Attention Pre- to Post-Supplement Intake at Week 12 | Pre- to 1 hour post- supplement intake at week 12 of the intervention.
  Assessed as the signal detection measure of a subject's sensitivity to the target sequence (A') during the Cambridge Neuropsychological Test Automated Battery rapid visual information processing test.

SECONDARY OUTCOMES:
Verbal Episodic Memory Performance at Week 4 | Week 4
  Assessed as the number of errors made on the Cambridge Neuropsychological Test Automated Battery verbal paired associates task.
Verbal Episodic Memory Performance at Week 8 | Week 8
  Assessed as the number of errors made on the Cambridge Neuropsychological Test Automated Battery verbal paired associates task
Verbal Episodic Memory Performance at Week 12 | Week 12
  Assessed as the number of errors made on the Cambridge Neuropsychological Test Automated Battery verbal paired associates task.
Working Memory Performance at Week 4 | Week 4
  Assessed as the longest sequence successfully completed during the Cambridge Neuropsychological Test Automated Battery digit span task.
Working Memory Performance at Week 8 | Week 8
  Assessed as the longest sequence successfully completed during the Cambridge Neuropsychological Test Automated Battery digit span task
Working Memory Performance at Week 12 | Week 12
  Assessed as the longest sequence successfully completed during the Cambridge Neuropsychological Test Automated Battery digit span task.
Spatial Planning and Working Memory Performance at Week 4 | Week 4
  Assessed as the number of problems completed using the minimum number of moves during the Cambridge Neuropsychological Test Automated Battery stockings of Cambridge task
Spatial Planning and Working Memory Performance at week 8 | Week 8
  Assessed as the number of problems completed using the minimum number of moves during the Cambridge Neuropsychological Test Automated Battery stockings of Cambridge task
Spatial Planning and Working Memory Performance at Week 12 | Week 12
  Assessed as the number of problems completed using the minimum number of moves during the Cambridge Neuropsychological Test Automated Battery stockings of Cambridge task.
Sustained Attention Performance at Week 4 | Week 4
  Assessed as the signal detection measure of a subject's sensitivity to the target sequence (A') during the Cambridge Neuropsychological Test Automated Battery rapid visual information processing test.
Sustained Attention Performance at week 8 | Week 8
  Assessed as the signal detection measure of a subject's sensitivity to the target sequence (A') during the Cambridge Neuropsychological Test Automated Battery rapid visual information processing test
Sustained Attention Performance at Week 12 | Week 12
  Assessed as the signal detection measure of a subject's sensitivity to the target sequence (A') during the Cambridge Neuropsychological Test Automated Battery rapid visual information processing test.
Subjective Memory Complaints at Week 4 | Week 4
  Assessed using the Everyday Memory Questionnaire - Revised. Retrieval subscale (seven items, range 0-28) and the attentional subscale (four items, score range 0-16). A higher score indicates greater presence of subjective memory or attention difficulties.
Subjective Memory Complaints at Week 8 | Week 8
  Assessed using the Everyday Memory Questionnaire - Revised. Retrieval subscale (seven items, range 0-28) and the attentional subscale (four items, score range 0-16). A higher score indicates greater presence of subjective memory or attention difficulties.
Subjective Memory Complaints at Week 12 | Week 12
  Assessed using the Everyday Memory Questionnaire - Revised. Retrieval subscale (seven items, range 0-28) and the attentional subscale (four items, score range 0-16). A higher score indicates greater presence of subjective memory or attention difficulties.
Self-reported Sleep Quality at Week 4 | Week 4
  Assessed using the Pittsburgh sleep quality index. Each component is scored from 0 to 3, to give a global score between 0 and 21.Higher scores signify poorer subjective sleep quality.
Self-reported Sleep Quality at Week 8 | Week 8
  Assessed using the Pittsburgh sleep quality index. Each component is scored from 0 to 3, to give a global score between 0 and 21. Higher scores signify poorer subjective sleep quality.
Self-reported Sleep Quality at Week 12 | Week 12
  Assessed using the Pittsburgh sleep quality index. Each component is scored from 0 to 3, to give a global score between 0 and 21. Higher scores signify poorer subjective sleep quality.
Self-reported Hot Flash Severity and Frequency at Week 4 | Week 4
  Assessed using the Hot flush rating scale. Split into two sub-sections: frequency and problem rating. Scored on a scale from 1 -10, the overall problem rating is calculated as the mean from the three items. A higher score indicates greater problem rating.
Self-reported Hot Flash Severity and Frequency at Week 8 | Week 8
  Assessed using the Hot flush rating scale. Split into two sub-sections: frequency and problem rating. Scored on a scale from 1 -10, the overall problem rating is calculated as the mean from the three items. A higher score indicates greater problem rating.
Self-reported Hot Flash Severity and Frequency at Week 12 | Week 12
  Assessed using the Hot flush rating scale. Split into two sub-sections: frequency and problem rating. Scored on a scale from 1 -10, the overall problem rating is calculated as the mean from the three items. A higher score indicates greater problem rating.
Anxiety Symptoms at Week 4 | Week 4
  Assessed using the anxiety sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe anxiety symptoms.
Anxiety Symptoms at Week 8 | Week 8
  Assessed using the anxiety sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe anxiety symptoms.
Anxiety Symptoms at Week 12 | Week 12
  Assessed using the anxiety sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe anxiety symptoms.
Stress symptoms at Week 4 | Week 4
  Assessed using the stress sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe stress symptoms.
Stress Symptoms at Week 8 | Week 8
  Assessed using the stress sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe stress symptoms.
Stress Symptoms at Week 12 | Week 12
  Assessed using the stress sub-scale of the Depression, Anxiety and stress scale - 21 items. Assessed on a scale from 0 - 3 over 7 questions, with a maximum score of 42. Higher scores indicate more severe stress symptoms.
Quality of Life Score at Week 4 | Week 4
  Assessed using the menopause specific quality of life questionnaire. The score for each domain ranges from 1 to 8, and the overall problem rating is calculated as the mean score. Higher score represents worse quality of life.
Quality of Life Score at Week 8 | Week 8
  Assessed using the menopause specific quality of life questionnaire. The score for each domain ranges from 1 to 8, and the overall problem rating is calculated as the mean score. Higher score represents worse quality of life.
Quality of Life Score at Week 12 | Week 12
  Assessed using the menopause specific quality of life questionnaire. The score for each domain ranges from 1 to 8, and the overall problem rating is calculated as the mean score. Higher score represents worse quality of life.
Change in Handgrip Strength from baseline to Week 12 | Baseline and Week 12
  Assessed using a handgrip dynamometer.
change in Leg Extensor Submaximal Strength from baseline to Week 12 | Baseline and Week 12
  Assessed using the 4-6RM leg extensor strength test.
Change in Isometric Mid-thigh Pull Strength from baseline to Week 12 | Baseline and Week 12
  Assessed using a portable back and leg dynamometer in a standing horizontal pull configuration
Change in the Number of Reps Completed in the 30 Second Sit-to-stand Test from baseline to week 12 | baseline and Week 12
  Assessed as the number of reps completed in 30 seconds
Change in Appendicular Lean Mass from baseline to Week 12 | Baseline and Week 12
  Measured using dual X-ray Absorptiometry
Felt-affect Visual Analogue score at week 4 | Week 4
  To assess the perceived impact of the supplement on mood and cognitive function. Higher scores indicate greater perceived impact
Felt-affect Visual Analogue score at week 8 | Week 8
  To assess the perceived impact of the supplement on mood and cognitive function. Higher scores indicate greater perceived impact
Felt-affect Visual Analogue score at week 12 | Week 12
  To assess the perceived impact of the supplement on mood and cognitive function. Higher scores indicate greater perceived impact
Exercise Enjoyment at week 1 | Week 1
  Assessed as overall score on the physical activity enjoyment scale on a likert scale from 1 to 7. Overall score is calculated as a sum of all scores once reverse items have been calculated. Higher scores indicate greater exercise enjoyment.
Exercise Enjoyment at week 4 | Week 4
  Assessed as overall score on the physical activity enjoyment scale on a likert scale from 1 to 7. Overall score is calculated as a sum of all scores once reverse items have been calculated. Higher scores indicate greater exercise enjoyment.
Exercise Enjoyment at week 8 | Week 8
  Assessed as overall score on the physical activity enjoyment scale on a likert scale from 1 to 7. Overall score is calculated as a sum of all scores once reverse items have been calculated. Higher scores indicate greater exercise enjoyment.
Exercise Enjoyment at week 12 | Week 12
  Assessed as overall score on the physical activity enjoyment scale on a likert scale from 1 to 7. Overall score is calculated as a sum of all scores once reverse items have been calculated. Higher scores indicate greater exercise enjoyment.
Change in Verbal Episodic Memory Performance from Pre- to Post-Supplement Intake in Week 1. | Pre- to 1 hour post- supplement intake in week 1
  Measured as the number of errors during the Cambridge Neuropsychological Test Automated Battery verbal Paired associates task.
Change in Verbal Episodic Memory Performance From Pre- to Post-Supplement Intake in Week 12 | Pre- to 1 hour post- supplement intake in week 12
  Measured as the number of errors during the Cambridge Neuropsychological Test Automated Battery verbal Paired associates task.
Change in Working Memory Performance From Pre- to Post-Supplement Intake in Week 1 | Pre- to 1 hour post- supplement intake in week 1
  Measured as the longest sequence successfully completed during the Cambridge Neuropsychological Test Automated Battery backwards digit span task.
Change In Working Memory Performance From Pre- to Post-Supplement Intake in Week 12. | Pre- to 1 hour post- supplement intake in week 12
  Measured as the longest sequence successfully completed during the Cambridge Neuropsychological Test Automated Battery backwards digit span task.
Change in Spatial Planning and Working Memory Performance From Pre- to Post-Supplement Intake in Week 1. | Pre- to 1 hour post- supplement intake in week 1.
  Measured as the number of problems completed using the minimum number of moves during the Cambridge Neuropsychological Test Automated Battery stockings of Cambridge task.
Change in Spatial Planning and Working Memory Performance From Pre- to Post-Supplement Intake in Week 1. | Pre- to 1 hour post- supplement intake in week 12
  Measured as the number of problems completed using the minimum number of moves during the Cambridge Neuropsychological Test Automated Battery stockings of Cambridge task.
Change in Mood State From Pre- to Post- Supplement Intake in week 1 | Pre- to 1 hour post- supplement intake in week 1.
  Assessed using the Bond-Lader visual analogue scale. Scores can be split into alertness, contentment and calmness with lower scores indicating a higher experience of the positive mood state.
Change in Mood State From Pre- to Post- Supplement Intake in Week 12 | Pre- to 1 hour post- supplement intake in week 12
  Assessed using the Bond-Lader visual analogue scale. Scores can be split into alertness, contentment and calmness with lower scores indicating a higher experience of the positive mood state.
Change in total body fat percentage from baseline to Week 12 | Baseline and Week 12
  Measured using dual X-ray Absorptiometry

OTHER OUTCOMES:
A Panel of Serum Steroid Hormones (e.g. Oestradiol, Progesterone, Testosterone and Cortisol) at Week 4 | Week 4
  Analysed using LCMS from a serum sample.
A Panel of Serum Steroid Hormones (e.g. Oestradiol, Progesterone, Testosterone and Cortisol) at Week 8 | Week 8
  Analysed using LCMS from a serum sample.
A Panel of Serum Steroid Hormones (e.g. Oestradiol, Progesterone, Testosterone and Cortisol) at Week 12 | Week 12
  Analysed using LCMS from a serum sample.
Brain Derived Neurotrophic Factor at week 4 | Week 4
  Analysed using ELISA from obtained serum sample
Brain Derived Neurotrophic Factor at Week 8 | Week 8
  Analysed using ELISA from obtained serum sample
Brain Derived Neurotrophic Factor at Week 12 | Week 12
  Analysed using ELISA from obtained serum sample
Change From Baseline in Monoamine Oxidase A & B Activity at Week 4 | Baseline to Week 4
  Analysed using Amplex assay kit.
Change from baseline in Monoamine oxidase A & B activity at week 8 | Baseline to week 8
  Analysed using Amplex assay kit.
Change from baseline in Monoamine oxidase A & B activity at week 12 | Baseline to week 12
  Analysed using Amplex assay kit.
Change from baseline in plasma sarmentosin at week 4 | Baseline to week 4
  Analysed using LCMS
Change from baseline in plasma sarmentosin at week 8 | Baseline to week 8
  Analysed using LCMS
Change from baseline in plasma sarmentosin at week 12 | Baseline to week 12
  Analysed using LCMS
Inflammatory Cytokines (IL6, TNF-α) at week 4 | Week 4
  Analysed using ELISA
Inflammatory cytokines (e.g. IL6, TNF-α) at week 8 | Week 8
  Analysed using ELISA
Inflammatory cytokines (e.g. IL6, TNF-α) at week 12 | Week 12
  Analysed using ELISA
Change in Sarmentosin Levels From Pre- to Post-Supplement Intake in Week 1. | Pre- to 1 hour post- supplement intake in week 1
  Analysed using LCMS
Change in Sarmentosin Levels From Pre- to Post-Supplement Intake in Week 12 | Pre- to 1 hour post- supplement intake in week 12
  Analysed using LCMS
Change in L-theanine Levels From Pre- to Post-Supplement Intake in Week 1. | Pre- to 1 hour post- supplement intake in week 1
  Analysed using LCMS
Change in L-theanine Levels From Pre- to Post-Supplement Intake in Week 12 | Pre- to 1 hour post- supplement intake in week 12
  Analysed using LCMS
Change in Plasma Monoamine Oxidase A and B Activity From Pre- to Post-Supplement Intake in Week 1 | Pre- to 1 hour post- supplement intake in week 1
  Analysed using amplex assay kits
Change in Plasma Monoamine Oxidase A and B Activity From Pre- to Post-Supplement Intake in Week 12 | Pre- to 1 hour post- supplement intake in week 12
  Analysed using amplex assay kits

CONTACTS AND LOCATIONS:
Locations (1):
- Carnegie School of Sport, Leeds, North Humberside, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided